CLINICAL TRIAL: NCT04762303
Title: Spread and Scale of a Polypharmacy App to Improve Health Outcomes of Older Adults Living in New Brunswick Nursing Homes: an Effectiveness-Implementation Hybrid Type 2 Study Design for a Stepped Wedge Cluster Randomized Trial
Brief Title: Spread and Scale of a Polypharmacy App
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Centre for Innovation and Research in Aging, Canada (Other)
Collaborators: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other); Horizon Health Network (Other); Missing Link Technologies (Unknown); New Brunswick Community College (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Supportive Care
Other Study IDs: C0061
Record Dates: First submitted 2021-02-09; First posted 2021-02-21 (Actual); Last update posted 2021-06-16 (Actual); Status verified 2021-02

CONDITIONS: Polypharmacy; Deprescribing; Adverse Drug Event
Keywords: Polypharmacy; Deprescribing; Adverse Drug Event; Older Adults; Long-Term Care; Medication Use; Medication Review; Nursing Home; Prescription Check-Up
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MedReviewRx (Experimental): During the intervention phase, MedReviewRx will be made available to nursing homes with the understanding that it will be used to facilitate medication reviews and prescription check-ups. MedReviewRx provides clinicians with access to individualized and prioritized deprescribing information from MedSafer which: a) identifies potentially inappropriate medications (PIMs), b) explains why the medication is potentially inappropriate and c) provides instructions on how to safely stop/taper the medication.
  Interventions: Other: MedReviewRx
- No MedReviewRx (No Intervention): During the control phase, MedReviewRx will not be accessible to health care professionals at the nursing homes. This serves to obtain baseline deprescribing levels for each nursing home.

INTERVENTIONS:
Other: MedReviewRx — During the intervention phase, MedReviewRx will be made available to nursing homes with the understanding that it will be used to facilitate medication reviews and prescription check-ups. MedReviewRx provides clinicians with access to individualized and prioritized deprescribing information from MedSafer which: a) identifies potentially inappropriate medications (PIMs), b) explains why the medication is potentially inappropriate and c) provides instructions on how to safely stop/taper the medication.
  Arms: MedReviewRx

SUMMARY:
Medication overload is an epidemic causing widespread harm, particularly to older Canadians. While most prescriptions are intended to help people live longer and healthier lives, taking multiple medications can increase frailty, and lead to dangerous side effects.This is a mixed-methods study to determine the impact of MedReviewRx on prescribing in New Brunswick Nursing Homes (NBNHs). MedReviewRx is an application which allows MedSafer to analyze a person's medications and medical conditions and produce a report with suggestions for how to simplify medications and make them safer. MedSafer reports will be used to assist physicians and pharmacists identify potentially inappropriate medications (PIMs) and conduct medication reviews in NBNHs. The prevalence of PIMs in NBNHs before MedReviewRx will be measured and the change in PIM use after implementation will be calculated. User experience with MedSafer reports and MedReviewRx will be explored. Patient and Family attitudes towards deprescribing will also be studied. Investigators hypothesize that implementing MedReviewRx in New Brunswick Nursing Homes (NBNHs) will promote deprescribing which will lead to a decrease in the number of PIMs and a decrease in medication costs for older adults living in NBNHs.

DETAILED DESCRIPTION:
Medication overload is an epidemic causing widespread harm, particularly to older Canadians. While most prescriptions are intended to help people live longer and healthier lives, taking multiple medications can increase frailty, and lead to dangerous side effects. As people age, the way medicines work may change and certain medicines are more likely cause problems with memory, thinking and balance. To minimize these risks, it is important to regularly review all medicines an older adult is taking. A medication review can be complicated, and it takes time. MedSafer is a computer program that helps physicians and pharmacists identify medicines that may no longer be needed or are dangerous. The software runs an analysis of a person's medications and medical conditions and produces a report with suggestions for how to simplify combinations of medications and make them safer. The process of safely reducing medications is called deprescribing. A computer application powered by MedSafer was built for nursing homes. This Polypharmacy App was piloted at a large urban nursing home. Initial impression of the system was positive. Improvements were made and it was rebranded as MedReviewRx. The current study will test MedReviewRx in other nursing homes in New Brunswick. MedReviewRx allows health care providers (prescribers, pharmacists and nurses) in nursing homes to access MedSafer analysis on a tablet or laptop. The investigators expect that access to this information will promote deprescribing in nursing homes, reduce potentially inappropriate medications (PIMs) and result in cost savings.

This study is a hybrid type 2 effectiveness-implementation design for quality improvement research that will make use of mixed methods of evaluation. Implementation consists of using MedReviewRx. Effectiveness analysis consists of measuring the impact of the MedReviewRx on PIMs. Exploratory surveys (the mixed methods component of the study) which look at qualitative and quantitative user feedback and patient and caregiver attitudes about deprescribing will be used to explain study findings. Informal feedback, surveys and semi-structured interviews will be used to examine user experience with MedReviewRx. The Revised Patient Attitude Towards Deprescribing (rPATD) questionnaire "older adult" version for the patients and a "caregiver" version for family members/substitute decision makers will be used to describe patient and family member attitudes about deprescribing medications.

Estimated study duration is 18 months. Deployment will approximate a Stepped Wedge Cluster Randomized Trial Design (SW-CRT). This type of study design allows us to approximate a randomized clinical trial. It has many advantages and is considered the most robust type of study design for a pragmatic quality improvement intervention. All clusters act as an internal control (before and after) as well as a control for the other clusters (external control). This novel study design addresses issues with seasonality and allows all clusters to participate in the intervention, which is an advantage when the intervention is related to quality improvement. It also allows us to measure for within and between cluster comparisons. Moreover, stepped-wedge trials are claimed by many researchers to have a statistical advantage over parallel cluster randomized trials. In the same direction, more researchers state that on one hand, for cluster randomized trials (CRTs), the stepped wedge design is far more efficient than the parallel group and ANCOVA design in terms of sample size. On the other hand, these researchers also state that the stepped wedge design requires a substantially smaller sample size than a parallel group and ANCOVA design.

The study will have three clusters with a combined total of approximately 750 nursing home beds. Nursing home resident turnover rates may be as high as 30% per year therefore the researchers anticipate that up to 1000 residents will be screened by MedSafer at least once and 300 of them, or more, will have a potentially inappropriate medication (PIM) identified. A random generator was used to place participating nursing homes into the following three clusters:

Cluster 1: 3 months control + 9 months intervention

Cluster 2: 6 months control + 6 months intervention

Cluster 3: 9 months control + 3 months intervention

As illustrated, the study will begin with a minimum three-month control phase. During the control phase, MedReviewRx will not be accessible to health care professionals at the nursing homes. This serves to obtain baseline deprescribing levels for each nursing home. Every three to four months thereafter, a cluster of nursing homes will enter intervention mode.

During the control phase, nursing home residents and their families or substitute decision makers will be recruited to complete a survey to explore patient attitudes about deprescribing in this NB study population. The rPATD questionnaire "older adult" version will be provided to nursing home residents and the "caregiver" version will be provided to family members and substitute decision makers. Survey questions will be entered in Lime survey to promote electronic completion whenever possible. A recruitment poster will be displayed at study sites and a recruitment communication will be sent to family members and substitute decision makers identified in the resident's admission package. Paper copies will also be available from the study site contact. Residents and family members who ask nursing home staff about the survey will have their contact information forwarded to the Centre for Innovation and Research in Aging (CIRA) research manager to answer questions and obtain verbal consent to have a survey e-mailed to them. If e-mail is not available, a research assistant will contact the participant to administer the survey over the phone. Study site contacts may also distribute paper copies of the surveys if requested and permitted by the study site. Stamped envelopes addressed to the CIRA research manager will be provided with each paper survey distributed.

Also during the control phase, health care providers and study site staff will be recruited to register for MedReviewRx. A recruitment communication will be sent by e-mail and placed in study site mailboxes. Study recruitment will also be encouraged at interdisciplinary nursing home meetings such as Pharmacy and Therapeutics and Medical Advisory Committee meetings. User training will be provided by the study site contact or designate(s) as determined by the site-specific implementation plan. Nursing home site contacts will participate in an interview to evaluate MedReviewRx implementation. Implementation interviews will be conducted within the first 3 months of the site intervention phase videoconference by the CIRA research manager or designate via telephone or Zoom.

During the intervention phase, MedReviewRx will be made available to nursing homes with the understanding that it will be used to facilitate medication reviews and prescription check-ups. MedReviewRx provides clinicians with access to individualized and prioritized deprescribing information from MedSafer which: a) identifies PIMs, b) explains why the medication is potentially inappropriate and c) provides instructions on how to safely stop/taper the medication. Nursing homes will also have the option to print MedSafer deprescribing reports from MedReviewRx for clinicians who do not have computer access or who choose not to register to use MedReviewRx. If reports are printed, they will be placed in a binder for the prescriber to sign and date indicating that they have read the report. Prescribers and nursing home staff will be encouraged to write feedback directly on the report if they wish too. To assess the proportion of reports that were read, and feedback provided on the reports, signed reports will be kept in a locked cabinet for research assistants to collect.

Clinicians will review deprescribing opportunities (electronically or via a paper report) and determine if medications can be tapered or stopped. Medication changes are discussed with the resident or substitute decision maker as part of usual care. This process will not change with the implementation of MedReviewRx. If the prescriber decides to alter a medication based on the deprescribing opportunities provided by MedSafer and their expert knowledge, the prescriber will do so in the same manner as they did prior to implementation of MedReviewRx, and discussion with the resident and/or substitute decision maker will occur according to the process in place at each nursing home. During the intervention phase, an analysis of deprescribing opportunities will be conducted by MedSafer once every 3 months for each resident in the nursing home. Results will be stored in the MedReviewRx system to be accessed at any time.

User feedback on MedReviewRx and MedSafer deprescribing information will be solicited from prescribers, pharmacists and nursing home staff throughout the study using surveys. Surveys may be completed via Lime Survey, on paper or by telephone (depending on the preference of the person). Three surveys will be distributed by e-mail to registered MedReviewRx users as well as other study site prescribers, pharmacists and nurses who may have access to printed reports from MedReviewRx. A MedReviewRx user feedback survey will be distributed at the end of the first and third quarter of the intervention and an acceptability and feasibility survey will be distributed at the end of the study. Informal feedback received by e-mail from users will be reviewed and actioned by the CIRA research manager or designate. E-mail feedback will be documented anonymously in an excel spreadsheet and reported to the study principle investigators within 1 week of receipt to determine if tasks need to be submitted to the technical team for software updates. Rapid cycle improvements in usability of the system and MedSafer output will be made based on survey results and informal feedback.

Informal feedback written on printed MedSafer reports will be documented in an excel spreadsheet and included in the analysis of qualitative feedback provided by survey and interview. Frequency of MedReviewRx use will be measured electronically by counting the number of times a user accesses their account. Overall experience with the research project will be evaluated using semi-structured interview conducted at the end of the intervention period.

ELIGIBILITY:
Inclusion Criteria:

* All residents of the participating New Brunswick nursing homes (NBNHs)
* All residents who are 65 years of age or older
* All residents who are taking a potentially inappropriate medication (as identified by MedSafer)

Exclusion Criteria:

* If both the patient and proxy are unable to complete the survey, the patient will be excluded from the survey component of the study.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2021-08-01 (Estimated); Primary Completion 2022-07-31 (Estimated); Study Completion 2022-10-31 (Estimated)

PRIMARY OUTCOMES:
Impact of MedReviewRx on the prevalence of potentially inappropriate medications (PIMs) in New Brunswick nursing homes (NBNHs). | Baseline to 3 months
  The impact on PIMs will be determined by the proportion of nursing home residents who have one or more PIMs reduced or stopped after the treating physician receives a MedSafer report

SECONDARY OUTCOMES:
Proportion of patients with one or more PIM reduced or stopped following each cycle. | 90-days following the first intervention cycle (9-months)
  Sustainability
Proportion of patients with one or more PIM reduced or stopped following each cycle. | 90-days following the second intervention cycle (6-months)
  Sustainability
Proportion of patients with one or more PIM reduced or stopped following each cycle. | 90-days following the third intervention cycle (3-months)
  Sustainability
Number of deaths | 90-days following the first intervention cycle (9-months)
  Safety data
Number of deaths | 90-days following the second intervention cycle (6-months)
  Safety data
Number of deaths | 90-days following the third intervention cycle (3-months)
  Safety data
Number of fractures | 90-days following the first intervention cycle (9-months)
  Safety data
Number of fractures | 90-days following the second intervention cycle (6-months)
  Safety data
Number of fractures | 90-days following the third intervention cycle (3-months)
  Safety data
Number of falls | 90-days following the first intervention cycle (9-months)
  Safety data
Number of falls | 90-days following the second intervention cycle (6-months)
  Safety data
Number of falls | 90-days following the third intervention cycle (3-months)
  Safety data
Number of restraints | 90-days following the first intervention cycle (9-months)
  Safety data
Number of restraints | 90-days following the second intervention cycle (6-months)
  Safety data
Number of restraints | 90-days following the third intervention cycle (3-months)
  Safety data
Number of transfers to the hospital | 90-days following the first intervention cycle (9-months)
  Safety data
Number of transfers to the hospital | 90-days following the second intervention cycle (6-months)
  Safety data
Number of transfers to the hospital | 90-days following the third intervention cycle (3-months)
  Safety data
Change in functional status based on interRAI activities of daily living (ADL) scores. | 90-days following the first intervention cycle (9-months)
  The ADL Hierarchy ranges from 0 (no impairment) to 6 (total dependence)
Change in functional status based on interRAI activities of daily living (ADL) scores. | 90-days following the second intervention cycle (6-months)
  The ADL Hierarchy ranges from 0 (no impairment) to 6 (total dependence)
Change in functional status based on interRAI activities of daily living (ADL) scores. | 90-days following the third intervention cycle (3-months)
  The ADL Hierarchy ranges from 0 (no impairment) to 6 (total dependence)
Number of participants with transfers out of the institution (return to independent living) | 90-days following the first intervention cycle (9-months)
  Safety data
Number of participants with transfers out of the institution (return to independent living) | 90-days following the second intervention cycle (6-months)
  Safety data
Number of participants with transfers out of the institution (return to independent living) | 90-days following the third intervention cycle (3-months)
  Safety data
Number of participants with episodes of delirium based on responses to questions in Section C of the interRAI LTCF assessment form | 90-days following the first intervention cycle (9-months)
  0 (Behavior not present), 1 (Behavior present, consistent with usual functioning), 2 (Behavior present, appears different from usual functioning)
Number of participants with episodes of delirium based on responses to questions in Section C of the interRAI LTCF assessment form | 90-days following the second intervention cycle (6-months)
  0 (Behavior not present), 1 (Behavior present, consistent with usual functioning), 2 (Behavior present, appears different from usual functioning)
Number of participants with episodes of delirium based on responses to questions in Section C of the interRAI LTCF assessment form | 90-days following the third intervention cycle (3-months)
  0 (Behavior not present), 1 (Behavior present, consistent with usual functioning), 2 (Behavior present, appears different from usual functioning)
Number of changes from baseline in composite safety data | 90-days following the first intervention cycle (9-months)
  Deaths, fractures, falls, use of restraints, transfers to hospital, pressure ulcers and stage, in-dwelling catheter use, change in functional status, transfers out of the institution, episodes of delirium.
Number of changes from baseline in composite safety data | 90-days following the second intervention cycle (6-months)
  Deaths, fractures, falls, use of restraints, transfers to hospital, pressure ulcers and stage, in-dwelling catheter use, change in functional status, transfers out of the institution, episodes of delirium.
Number of changes from baseline in composite safety data | 90-days following the third intervention cycle (3-months)
  Deaths, fractures, falls, use of restraints, transfers to hospital, pressure ulcers and stage, in-dwelling catheter use, change in functional status, transfers out of the institution, episodes of delirium.
User experience with MedSafer reports and MedReviewRx. Measured by survey responses. | 90-days following the first intervention cycle (9-months)
  Open ended questions, multiple choice questions and Likert scales: 1 (not at all) to 10 (very much), strongly disagree to strongly agree, very unlikely to very likely.
User experience with MedSafer reports and MedReviewRx. Measured by survey responses. | 90-days following the second intervention cycle (6-months)
  Open ended questions, multiple choice questions and Likert scales: 1 (not at all) to 10 (very much), strongly disagree to strongly agree, very unlikely to very likely.
User experience with MedSafer reports and MedReviewRx. Measured by survey responses. | 90-days following the third intervention cycle (3-months)
  Open ended questions, multiple choice questions and Likert scales: 1 (not at all) to 10 (very much), strongly disagree to strongly agree, very unlikely to very likely.
User experience with MedSafer reports and MedReviewRx. Measured through interview data. | 90-days following the first intervention cycle (9-months)
  Open ended questions
User experience with MedSafer reports and MedReviewRx. Measured through interview data. | 90-days following the second intervention cycle (6-months)
  Open ended questions
User experience with MedSafer reports and MedReviewRx. Measured through interview data. | 90-days following the third intervention cycle (3-months)
  Open ended questions
User experience with MedSafer reports and MedReviewRx. Measured through informal feedback received by the study team. | 90-days following the first intervention cycle (9-months)
  Operationalizing testing
User experience with MedSafer reports and MedReviewRx. Measured through informal feedback received by the study team. | 90-days following the second intervention cycle (6-months)
  Operationalizing testing
User experience with MedSafer reports and MedReviewRx. Measured through informal feedback received by the study team. | 90-days following the third intervention cycle (3-months)
  Operationalizing testing

OTHER OUTCOMES:
Cost savings | 1 year
  Cost savings analysis related to cost saved from medications (actual price of the medication as well as dispensing fees) balanced with the cost of deployment of MedSafer including maintaining the program with updates and user support.
Patient and family attitudes about deprescribing | 90-days following the first intervention cycle (9-months)
  Patient and family attitudes about deprescribing will be reported using survey responses collected from the revised Patient Attitude Towards Deprescribing (rPATD) questionnaires. Questionnaires contain 19 questions (caregiver version) and 22 questions (older adult version) with answers ranging from "strongly agree" to strongly disagree".
Patient and family attitudes about deprescribing | 90-days following the second intervention cycle (6-months)
  Patient and family attitudes about deprescribing will be reported using survey responses collected from the revised Patient Attitude Towards Deprescribing (rPATD) questionnaires. Questionnaires contain 19 questions (caregiver version) and 22 questions (older adult version) with answers ranging from "strongly agree" to strongly disagree".
Patient and family attitudes about deprescribing | 90-days following the third intervention cycle (3-months)
  Patient and family attitudes about deprescribing will be reported using survey responses collected from the revised Patient Attitude Towards Deprescribing (rPATD) questionnaires. Questionnaires contain 19 questions (caregiver version) and 22 questions (older adult version) with answers ranging from "strongly agree" to strongly disagree".

CONTACTS AND LOCATIONS:
Overall Officials: Carole Goodine, Pharm D, Principal Investigator — Horizon Health Network; Emily McDonald, MD, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre
Locations (5):
- Canada (5):
  - York Care Centre, Fredericton, New Brunswick
  - Faubourg du Mascaret, Moncton, New Brunswick
  - Spencer Nursing Home, Moncton, New Brunswick
  - Shannex Embassy Hall, Quispamsis, New Brunswick
  - Loch Lomond Villa, Saint John, New Brunswick

IPD SHARING:
Plan to Share IPD: Yes
Non-pharma academic researchers may contact the principal investigator by email one year following the primary publication for access to data which will be shared via password-protected excel document.
Supporting Information: Study Protocol
Time Frame: Made available for 1 year following the publication of the primary manuscript from the trial.
Access Criteria: Contact study primary investigators at emily.mcdonald@mcgill.ca or Carole.goodine@horizonnb.ca

REFERENCES:
- [Background] AlRasheed MM, Alhawassi TM, Alanazi A, Aloudah N, Khurshid F, Alsultan M. Knowledge and willingness of physicians about deprescribing among older patients: a qualitative study. Clin Interv Aging. 2018 Aug 6;13:1401-1408. doi: 10.2147/CIA.S165588. eCollection 2018. PMID 30122912
- [Background] Caputo A. Trends of psychology-related research on euthanasia: a qualitative software-based thematic analysis of journal abstracts. Psychol Health Med. 2015;20(7):858-69. doi: 10.1080/13548506.2014.993405. Epub 2014 Dec 20. PMID 25530297
- [Background] Brath H, Mehta N, Savage RD, Gill SS, Wu W, Bronskill SE, Zhu L, Gurwitz JH, Rochon PA. What Is Known About Preventing, Detecting, and Reversing Prescribing Cascades: A Scoping Review. J Am Geriatr Soc. 2018 Nov;66(11):2079-2085. doi: 10.1111/jgs.15543. Epub 2018 Oct 18. PMID 30335185
- [Background] Conklin J, Farrell B, Suleman S. Implementing deprescribing guidelines into frontline practice: Barriers and facilitators. Res Social Adm Pharm. 2019 Jun;15(6):796-800. doi: 10.1016/j.sapharm.2018.08.012. Epub 2018 Sep 18. PMID 30241874
- [Background] Dills H, Shah K, Messinger-Rapport B, Bradford K, Syed Q. Deprescribing Medications for Chronic Diseases Management in Primary Care Settings: A Systematic Review of Randomized Controlled Trials. J Am Med Dir Assoc. 2018 Nov;19(11):923-935.e2. doi: 10.1016/j.jamda.2018.06.021. Epub 2018 Aug 11. PMID 30108032
- [Background] Djatche L, Lee S, Singer D, Hegarty SE, Lombardi M, Maio V. How confident are physicians in deprescribing for the elderly and what barriers prevent deprescribing? J Clin Pharm Ther. 2018 Aug;43(4):550-555. doi: 10.1111/jcpt.12688. Epub 2018 Apr 22. PMID 29682764
- [Background] McDonald EG, Wu PE, Rashidi B, Forster AJ, Huang A, Pilote L, Papillon-Ferland L, Bonnici A, Tamblyn R, Whitty R, Porter S, Battu K, Downar J, Lee TC. The MedSafer Study: A Controlled Trial of an Electronic Decision Support Tool for Deprescribing in Acute Care. J Am Geriatr Soc. 2019 Sep;67(9):1843-1850. doi: 10.1111/jgs.16040. Epub 2019 Jun 27. PMID 31250427
- [Background] Sirois C, Ouellet N, Reeve E. Community-dwelling older people's attitudes towards deprescribing in Canada. Res Social Adm Pharm. 2017 Jul-Aug;13(4):864-870. doi: 10.1016/j.sapharm.2016.08.006. Epub 2016 Aug 31. PMID 27663392
- [Background] Thillainadesan J, Gnjidic D, Green S, Hilmer SN. Impact of Deprescribing Interventions in Older Hospitalised Patients on Prescribing and Clinical Outcomes: A Systematic Review of Randomised Trials. Drugs Aging. 2018 Apr;35(4):303-319. doi: 10.1007/s40266-018-0536-4. PMID 29541966
- [Background] van der Sluijs R, Fiddelers AAA, Waalwijk JF, Reitsma JB, Dirx MJ, den Hartog D, Evers SMAA, Goslings JC, Hoogeveen WM, Lansink KW, Leenen LPH, van Heijl M, Poeze M. The impact of the Trauma Triage App on pre-hospital trauma triage: design and protocol of the stepped-wedge, cluster-randomized TESLA trial. Diagn Progn Res. 2020 Jun 18;4:10. doi: 10.1186/s41512-020-00076-1. eCollection 2020. PMID 32566758
- [Background] Barker D, D'Este C, Campbell MJ, McElduff P. Minimum number of clusters and comparison of analysis methods for cross sectional stepped wedge cluster randomised trials with binary outcomes: A simulation study. Trials. 2017 Mar 9;18(1):119. doi: 10.1186/s13063-017-1862-2. PMID 28279222
- [Background] Woertman W, de Hoop E, Moerbeek M, Zuidema SU, Gerritsen DL, Teerenstra S. Stepped wedge designs could reduce the required sample size in cluster randomized trials. J Clin Epidemiol. 2013 Jul;66(7):752-8. doi: 10.1016/j.jclinepi.2013.01.009. Epub 2013 Mar 22. PMID 23523551
- [Background] Kim J, Parish AL. Polypharmacy and Medication Management in Older Adults. Nurs Clin North Am. 2017 Sep;52(3):457-468. doi: 10.1016/j.cnur.2017.04.007. PMID 28779826
- [Background] Lavan AH, Gallagher P. Predicting risk of adverse drug reactions in older adults. Ther Adv Drug Saf. 2016 Feb;7(1):11-22. doi: 10.1177/2042098615615472. PMID 26834959
- [Background] By the American Geriatrics Society 2015 Beers Criteria Update Expert Panel. American Geriatrics Society 2015 Updated Beers Criteria for Potentially Inappropriate Medication Use in Older Adults. J Am Geriatr Soc. 2015 Nov;63(11):2227-46. doi: 10.1111/jgs.13702. Epub 2015 Oct 8. PMID 26446832
- [Background] O'Mahony D, O'Sullivan D, Byrne S, O'Connor MN, Ryan C, Gallagher P. STOPP/START criteria for potentially inappropriate prescribing in older people: version 2. Age Ageing. 2015 Mar;44(2):213-8. doi: 10.1093/ageing/afu145. Epub 2014 Oct 16. PMID 25324330
- [Background] Gallagher P, Barry P, O'Mahony D. Inappropriate prescribing in the elderly. J Clin Pharm Ther. 2007 Apr;32(2):113-21. doi: 10.1111/j.1365-2710.2007.00793.x. PMID 17381661
- [Background] Gutierrez-Valencia M, Izquierdo M, Cesari M, Casas-Herrero A, Inzitari M, Martinez-Velilla N. The relationship between frailty and polypharmacy in older people: A systematic review. Br J Clin Pharmacol. 2018 Jul;84(7):1432-1444. doi: 10.1111/bcp.13590. Epub 2018 May 3. PMID 29575094
- [Background] Thompson W, Farrell B. Deprescribing: what is it and what does the evidence tell us? Can J Hosp Pharm. 2013 May;66(3):201-2. doi: 10.4212/cjhp.v66i3.1261. No abstract available. PMID 23814291
- [Background] Hemming K, Kasza J, Hooper R, Forbes A, Taljaard M. A tutorial on sample size calculation for multiple-period cluster randomized parallel, cross-over and stepped-wedge trials using the Shiny CRT Calculator. Int J Epidemiol. 2020 Jun 1;49(3):979-995. doi: 10.1093/ije/dyz237. PMID 32087011
- [Background] Kim H, Park YH, Jung YI, Choi H, Lee S, Kim GS, Yang DW, Paik MC, Lee TJ. Evaluation of a technology-enhanced integrated care model for frail older persons: protocol of the SPEC study, a stepped-wedge cluster randomized trial in nursing homes. BMC Geriatr. 2017 Apr 18;17(1):88. doi: 10.1186/s12877-017-0459-7. PMID 28420324
- [Derived] McDonald EG, Estey JL, Davenport C, Bortolussi-Courval E, Gaudet J, Wilson Registe PP, Lee TC, Goodine C. Electronic Decision Support for Deprescribing in Older Adults Living in Long-Term Care: A Stepped-Wedge Cluster Randomized Trial. JAMA Netw Open. 2025 May 1;8(5):e2512931. doi: 10.1001/jamanetworkopen.2025.12931. PMID 40445620
- [Derived] Nadeau ME, Henry JL, Lee TC, Bortolussi-Courval E, Goodine C, McDonald EG. Spread and scale of an electronic deprescribing software to improve health outcomes of older adults living in nursing homes: study protocol for a stepped wedge cluster randomized trial. Trials. 2021 Nov 2;22(1):763. doi: 10.1186/s13063-021-05729-0. PMID 34727956